CLINICAL TRIAL: NCT02248350
Title: An Exercise Intervention to Mitigate Side-Effects Related to Androgen Deprivation Therapy Among Prostate Cancer Survivors.
Brief Title: An Exercise Intervention for Prostate Cancer Patients Receiving Androgen Deprivation Therapy
Acronym: MIGHTY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Georgetown_University_MC
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2016-07

CONDITIONS: Prostate Cancer; Physical Activity; Side-effects
Keywords: prostate cancer; physical activity; exercise; intervention; side effects; androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Group (Experimental): 8-weeks of supervised and home based exercise intervention, 3 times a week, 50-minutes a session for a total of 150/minutes a week
  Interventions: Behavioral: Supervised and Home Based Exercise
- Stretching Control group (Active Comparator): Informational booklet containing stretching exercises (20-minutes a day)
  Interventions: Behavioral: Stretching Control Group

INTERVENTIONS:
Behavioral: Supervised and Home Based Exercise — Participants will come to our community based research office for up to 50 min/session, 3-days/week of supervised exercise for 8-weeks. The exercise intensity will be tailored between 60-80% of their VO2max, as determined during baseline testing and with a rating of perceived exertion (RPE) of 11-14 on the 20-point scale.
  Arms: Exercise Group
Behavioral: Stretching Control Group — Participants randomized into the control group will be provided an informational booklet with stretching techniques and exercises and will be asked to stretch at least 20-minutes a day for the duration of the study.
  Arms: Stretching Control group

SUMMARY:
This main purpose of this study is to examine the effects of an exercise intervention to counteract adverse side effects related to Androgen Deprivation Therapy (ADT) in prostate cancer patients. Specifically, a supervised and home-based exercise program will be used to assess its impact on clinical and behavioral variables related to ADT in prostate cancer patients.

DETAILED DESCRIPTION:
This study will assess the feasibility of an exercise intervention to counteract adverse side effects related to ADT in prostate cancer (PCa) patients. Specifically, we will use an exercise intervention and assess its impact on bone mass density, Body Mass Index (BMI), hip/waist circumference levels, biomarkers (i.e., glucose, lipids), step count, grip strength, and health-related quality of life (HRQOL) using the Patient Reported Outcomes Measurement Information System (PROMIS®). In this 8-week two-arm randomized clinical trial, 40 PCa patients receiving ADT will be randomly assigned to an exercise (n=20) or a stretching control group (n=20) with a follow-up at 8-weeks.

ELIGIBILITY:
Inclusion Criteria:

* (1) Caucasian or African-American/Black men; (2) histologically confirmed non-metastatic PCa; (3) receiving ADT treatment for 9-months or less upon recruitment (and continue to receive treatment during the duration of the study); (4) 40 to 75 years old; (5) sedentary defined as <60 minutes of recreation or work requiring modest PA/week; (6) ability to perform the level of physical activity assessed by the Physical Activity Readiness Questionnaire (PAR-Q); (6) has access to a smartphone or computer with internet capabilities

Exclusion Criteria:

* (1) severe cardiac disease; (2) recent myocardial infarction; (3) treated for any other cancer; (4) any physical, psychological illness, and/or medical problems that restricted them from exercise; (5) and not willing or able to follow procedures specified by the study and/or instructions of the researcher.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | 8-weeks
  BMD will be measured by a DXA scan

SECONDARY OUTCOMES:
Physical Fitness | 8-weeks
  . The Bruce treadmill protocol will be used to examine VO2max using a ParvoMedics TrueOne 2400 metabolic cart
Muscle strength | 8-weeks
  Grip strength will be measured in a standardized way (three times in each arm) using a Jamar Dynamometer
Step Count | 8-weeks
  The Fit Bit reliably measures daily steps taken, distance walked, calories burned, and overall activity level.
Quality of Life (HRQOL) | 8-weeks
  The 10-item PROMIS® Global Health Scale will be used to assess key HRQOL domains including pain, fatigue, mental health, physical health, social health, and overall health
Hip/Waist Circumference | 8-weeks
  Anthropometric measures
Body Mass Index (BMI) | 8-weeks
  BMI will be measured according to height and weight
Glucose/Lipid levels | 8-weeks
  A fasting finger stick sample of blood (35 μl) will be assessed for immediate analysis of lipid panel (i.e., total cholesterol, HDL cholesterol, LDL cholesterol, VLDL cholesterol, triglycerides) and fasting glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Office of Minority Health and Health Disparities Research, Washington D.C., District of Columbia, United States